CLINICAL TRIAL: NCT01085136
Title: Phase III Randomized Trial of BIBW 2992 Plus Weekly Paclitaxel Versus Investigator's Choice of Chemotherapy Following BIBW 2992 Monotherapy in Non-small Cell Lung Cancer Patients Failing Previous Erlotinib or Gefitinib Treatment (LUX Lung 5)
Brief Title: LUX-Lung 5: Afatinib Plus Weekly Paclitaxel Versus Investigator's Choice of Single Agent Chemotherapy Following Afatinib Monotherapy in Non-small Cell Lung Cancer Patients Failing Erlotinib or Gefitinib
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.42; 2009-014563-39 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-03-10; First posted 2010-03-11 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

ARMS (2):
- Investigator's choice of chemotherapy (Active Comparator): Patients will be treated with investigator's choice of chemotherapy
  Interventions: Drug: Investigator´s choice of chemotherapy
- BIBW 2992 and Paclitaxel (Experimental): Patients will be treated with BIBW 2992daily with a medium dose and weekly administration of Paclitaxel at a dose of 80 mg/m2
  Interventions: Drug: BIBW 2992

INTERVENTIONS:
Drug: Investigator´s choice of chemotherapy — BIBW 2992 in a medium dose in combination with Paclitaxel to explore safety and efficacy versus investigator´s choice of chemotherapy
  Arms: Investigator's choice of chemotherapy
Drug: BIBW 2992 — BIBW 2992 will be given in a medium dose in combination with Paclitaxel to explore safety and efficacy versus investigator´s choice of chemotherapy
  Arms: BIBW 2992 and Paclitaxel

SUMMARY:
The primary objective of this randomized, open-label, active-controlled, multi-center trial is to determine the efficacy of BIBW 2992 given as an add-on to chemotherapy in patients with NSCLC Stage IIIb or IV progressing after BIBW 2992 monotherapy compared to chemotherapy alone in this patient population. Patients on both treatment arms will receive best supportive care in addition to study treatment. Patients enrolled into the trial will be treated and followed until death or lost to follow-up. Additional information on the health-related quality of life (HRQOL) will be collected.

ELIGIBILITY:
Inclusion criteria:

Part A

1. Patients with pathologically confirmed diagnosis of NSCLC Stage IIIB (with cytologically proven pleural effusion or pericardial effusion) or Stage IV who have failed treatment with erlotinib (Tarceva) or gefitinib (Iressa).
2. Patients should have received and failed at least one line of cytotoxic chemotherapy including a platinum-based regimen in patients eligible for platinum-based therapy and pemetrexed in pemetrexed eligible patients (unless pemetrexed is not considered a regulatory or clinical standard of care e.g. no label indication, no availability or no coverage by 3rd party payer(s)) for advanced or metastatic disease and have progressive disease following at least 12 weeks of treatment with erlotinib or gefitinib
3. Patients pretreated with taxane-based chemotherapy for advanced or metastatic disease must have experienced stable disease, partial or complete response as best response
4. Eastern Cooperative Oncology Group performance Score 0 or 1.
5. Patients with at least one tumor lesion that can accurately be measured by magnetic resonance imaging (MRI), or computed tomography (CT) in at least one dimension with longest diameter to be recorded as 10 mm but no less than double the slice thickness according to RESIST 1.1.
6. Male and female patients no less than 18 years of age.
7. Life expectancy of at least three (3) months.
8. Written informed consent that is consistent with ICH-GCP guidelines. Part B 1) Clinical benefit (disease stabilization or antitumor response) of 12 weeks duration in Part A of the trial determined on the second tumour assessment.

2.) Patients should have progressed in Part A according to RECIST 1.1 3.) New informed consent, including consent to biomarker sampling, must be signed before patients enter Part B of the trial

Exclusion criteria:

1. Previous treatment with BIBW 2992
2. Chemo-, hormone- (other than megestrol acetate, steroids required for maintenance non-cancer therapy or as premedication before chemotherapy) or immunotherapy within the past 4 weeks; except for TKI pretreatment (2 weeks only)
3. Active/symptomatic brain metastases including leptomeningeal disease. Patients with a history of treated brain metastasis must have a stable or normal brain MRT/CT scan at screening and be at least 4 weeks post-radiation or surgery for brain metastasis. Dexamethasone therapy will be allowed if administered as a stable dose for at least one month before randomization.
4. Significant or recent acute gastrointestinal disorders with diarrhea as a major symptom e.g., Crohn's disease, mal-absorption, or CTCAE Grade >2 diarrhea of any etiology at baseline
5. Patients who have any other life-threatening illness or organ system dysfunction, which in the opinion of the Investigator, would either compromise patient safety or interfere with the evaluation of the safety of the test drug
6. Other malignancies diagnosed within the past five (5) years (other than non-melanomatous skin cancer and in situ cervical cancer)
7. Radiotherapy within the past 2 weeks prior to treatment with the trial drug
8. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New york Heart Association (NYHA) functional classification of 3, unstable angina, or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to entering the trial.
9. Cardiac left ventricular function with resting ejection fraction of less than 50% measured by multigated blood pool imaging of the heart (MUGA scan) or echocardiogram .
10. Prior treatment with anthracyclines with a cumulative dose of doxorubicin (or equivalent) at or greater than 400 mg/m2
11. Absolute neutrophil count (ANC) at or less than 1500 / mm3
12. Platelet count at or less than 100,000 / mm3
13. Bilirubin at or greater than 1.5 mg / dL (>26 mol / L, SI unit equivalent)
14. Aspartate amino transferase (AST) or alanine amino transferase (ALT) at or greater than three times the upper limit of normal (if related to liver metastases at or greater than five times the upper limit of normal)
15. Serum creatinine at or greater 1.5 times the upper normal limit or calculated/measured creatinine clearance at or less than 45 mL/min
16. Women of child-bearing potential or men who are able to father a child unwilling to use a medically acceptable method of contraception during the trial
17. Pregnancy or breast feeding
18. Patients unable to comply with the protocol
19. Patients with any serious active infection including known human immunodeficiency virus (HIV), active hepatitis B or active hepatitis C
20. Known or suspected active drug or alcohol abuse
21. Pre-existing or current Interstitial lung disease (ILD) 22.)
22. Peripheral polyneuropathy of > Grade 2
23. Requirement for treatment with any of the pohibited concomitant medication listed in section 4.2.2.1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1154 (Actual)
Dates: Start 2010-02; Primary Completion 2013-10 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (97):
- Boehringer Ingelheim Investigational Site, Buenos Aires, Argentina
- Australia (5):
  - Boehringer Ingelheim Investigational Site, Kingswood, New South Wales
  - Boehringer Ingelheim Investigational Site, South Brisbane, Queensland
  - Boehringer Ingelheim Investigational Site, Box Hill, Victoria
  - Boehringer Ingelheim Investigational Site, Fitzroy, Victoria
  - Boehringer Ingelheim Investigational Site, Wodonga, Victoria
- Boehringer Ingelheim Investigational Site, Salzburg, Austria
- Belgium (7):
  - Boehringer Ingelheim Investigational Site, Aalst
  - Boehringer Ingelheim Investigational Site, Brussels
  - Boehringer Ingelheim Investigational Site, Duffel
  - Boehringer Ingelheim Investigational Site, La Louvière
  - Boehringer Ingelheim Investigational Site, Liège
  - Boehringer Ingelheim Investigational Site, Middelheim
  - Boehringer Ingelheim Investigational Site, Ottignies
- Boehringer Ingelheim Investigational Site, Porto Alegre, Brazil
- China (8):
  - Boehringer Ingelheim Investigational Site, Beijing
  - Boehringer Ingelheim Investigational Site, Changchun
  - Boehringer Ingelheim Investigational Site, Chengdu
  - Boehringer Ingelheim Investigational Site, Fuzhou
  - Boehringer Ingelheim Investigational Site, Guangzhou
  - Boehringer Ingelheim Investigational Site, Hangzhou
  - Boehringer Ingelheim Investigational Site, Nanjing
  - Boehringer Ingelheim Investigational Site, Shanghai
- Boehringer Ingelheim Investigational Site, Helsinki, Finland
- France (8):
  - Boehringer Ingelheim Investigational Site, Bayonne
  - Boehringer Ingelheim Investigational Site, Caen
  - Boehringer Ingelheim Investigational Site, Dijon
  - Boehringer Ingelheim Investigational Site, La Tronche
  - Boehringer Ingelheim Investigational Site, Lyon
  - Boehringer Ingelheim Investigational Site, Paris
  - Boehringer Ingelheim Investigational Site, Saint-Herblain
  - Boehringer Ingelheim Investigational Site, Villejuif
- Germany (9):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Essen
  - Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - Boehringer Ingelheim Investigational Site, Gauting
  - Boehringer Ingelheim Investigational Site, Hamburg
  - Boehringer Ingelheim Investigational Site, Hanover
  - Boehringer Ingelheim Investigational Site, Heidelberg
  - Boehringer Ingelheim Investigational Site, Mainz
  - Boehringer Ingelheim Investigational Site, Münster
- Hungary (3):
  - Boehringer Ingelheim Investigational Site, Budapest
  - Boehringer Ingelheim Investigational Site, Pécs
  - Boehringer Ingelheim Investigational Site, Törökbálint
- India (5):
  - Boehringer Ingelheim Investigational Site, Chennai
  - Boehringer Ingelheim Investigational Site, Jaipur
  - Boehringer Ingelheim Investigational Site, Maharashtra
  - Boehringer Ingelheim Investigational Site, Mumbai
  - Boehringer Ingelheim Investigational Site, Nashik, Maharashtra
- Israel (3):
  - Boehringer Ingelheim Investigational Site, Kfar Saba
  - Boehringer Ingelheim Investigational Site, Petah Tikva
  - Boehringer Ingelheim Investigational Site, Tel Litwinsky
- Italy (8):
  - Boehringer Ingelheim Investigational Site, Avellino
  - Boehringer Ingelheim Investigational Site, Aviano (PN)
  - Boehringer Ingelheim Investigational Site, Bergamo
  - Boehringer Ingelheim Investigational Site, Genova
  - Boehringer Ingelheim Investigational Site, Milan
  - Boehringer Ingelheim Investigational Site, Monza (mi)
  - Boehringer Ingelheim Investigational Site, Ravenna
  - Boehringer Ingelheim Investigational Site, Roma
- Boehringer Ingelheim Investigational Site, Distrito Federal, Mexico
- Netherlands (2):
  - Boehringer Ingelheim Investigational Site, Maastricht
  - Boehringer Ingelheim Investigational Site, Nieuwegein
- Peru (2):
  - Boehringer Ingelheim Investigational Site, Arequipa
  - Boehringer Ingelheim Investigational Site, La Victoria
- Poland (4):
  - Boehringer Ingelheim Investigational Site, Gdansk
  - Boehringer Ingelheim Investigational Site, Olsztyn
  - Boehringer Ingelheim Investigational Site, Otwock
  - Boehringer Ingelheim Investigational Site, Warsaw
- Russia (2):
  - Boehringer Ingelheim Investigational Site, Obninsk
  - Boehringer Ingelheim Investigational Site, Saint Petersburg
- South Korea (3):
  - Boehringer Ingelheim Investigational Site, Goyang
  - Boehringer Ingelheim Investigational Site, Hwasun
  - Boehringer Ingelheim Investigational Site, Seoul
- Spain (6):
  - Boehringer Ingelheim Investigational Site, A Coruña
  - Boehringer Ingelheim Investigational Site, Barcelona
  - Boehringer Ingelheim Investigational Site, Madrid
  - Boehringer Ingelheim Investigational Site, Mataró
  - Boehringer Ingelheim Investigational Site, Málaga
  - Boehringer Ingelheim Investigational Site, Valencia
- Taiwan (5):
  - Boehringer Ingelheim Investigational Site, Kaohsiung City
  - Boehringer Ingelheim Investigational Site, Taichung
  - Boehringer Ingelheim Investigational Site, Tainan
  - Boehringer Ingelheim Investigational Site, Taipei
  - Boehringer Ingelheim Investigational Site, Taoyuan District
- Ukraine (4):
  - Boehringer Ingelheim Investigational Site, Dnipropetrovks
  - Boehringer Ingelheim Investigational Site, Donetsk
  - Boehringer Ingelheim Investigational Site, Kharkiv
  - Boehringer Ingelheim Investigational Site, Kyiv
- United Kingdom (8):
  - Boehringer Ingelheim Investigational Site, Brighton
  - Boehringer Ingelheim Investigational Site, Dundee
  - Boehringer Ingelheim Investigational Site, Exeter
  - Boehringer Ingelheim Investigational Site, London
  - Boehringer Ingelheim Investigational Site, Maidstone
  - Boehringer Ingelheim Investigational Site, Manchester
  - Boehringer Ingelheim Investigational Site, Sutton, Surrey
  - Boehringer Ingelheim Investigational Site, Truro, Cornwall

REFERENCES:
- [Derived] Schuler M, Yang JC, Park K, Kim JH, Bennouna J, Chen YM, Chouaid C, De Marinis F, Feng JF, Grossi F, Kim DW, Liu X, Lu S, Strausz J, Vinnyk Y, Wiewrodt R, Zhou C, Wang B, Chand VK, Planchard D; LUX-Lung 5 Investigators. Afatinib beyond progression in patients with non-small-cell lung cancer following chemotherapy, erlotinib/gefitinib and afatinib: phase III randomized LUX-Lung 5 trial. Ann Oncol. 2016 Mar;27(3):417-23. doi: 10.1093/annonc/mdv597. Epub 2015 Dec 8. PMID 26646759

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PD = Progression Disease
Groups:
- Afatinib Monotherapy (Part A): Afatinib 50 mg film-coated tablet was orally administered once daily of each 28-day treatment course, with dose reductions to 40 mg/day and 30 mg/day (following the protocol-defined dose reduction scheme).
- Afatinib Plus Paclitaxel (Part B): Afatinib 40 mg film-coated tablet dose was orally administered once daily of each 28-day treatment course, with dose reductions to 30 mg/day and 20 mg/day (following the protocol defined dose reduction scheme) plus paclitaxel 80 mg/m2 administered via intravenous infusion once weekly (7 weeks on/1 week off; 2 dose reductions were allowed following the protocol defined dose reduction scheme and the current local summary of product characteristics).
- Investigators Choice of Chemotherapy (Part B): Reference therapy for Part B dose: Depending on schedule Intravenous or oral administration (2 dose reductions were allowed following the protocol defined dose reduction scheme and the current local summary of product characteristics).
Period: Part A
Arm/Group | Afatinib Monotherapy (Part A) | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Started | 1154 | 0 (Only Afatinib monotherapy administered in Part A) | 0
Randomized to Part B | 206 (Discontinued Part A -Randomized to Part B) | 0 | 0
Completed | 831 (Randomized to Part B & completed trial as per protocol, had PD, clinical progression.) | 0 | 0
Not Completed | 323 | 0 | 0
Not completed — Other Adverse event | 223 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0
Not completed — Refusal to continue trial medication | 64 | 0 | 0
Not completed — Other reason not defined above | 30 | 0 | 0
Period: Part B
Arm/Group | Afatinib Monotherapy (Part A) | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Started | 0 (Afatinib monotherapy not administered in Part B) | 138 | 68
Completed | 0 (Afatinib monotherapy not administered in Part B) | 87 (Completed trial as per protocol, had progressive disease, clinical signs or symptoms of progression) | 42 (Completed trial as per protocol, had progressive disease, clinical signs or symptoms of progression)
Not Completed | 0 | 51 | 26
Not completed — Other AE | 0 | 29 | 8
Not completed — Refusal to continue trial medication | 0 | 12 | 7
Not completed — Not treated | 0 | 4 | 8
Not completed — Other reason not defined above | 0 | 6 | 3

BASELINE CHARACTERISTICS:
Population: Treated set, i.e. all patients who were documented to have taken at least 1 dose of afatinib 50 mg in Part A of the trial and all patients who received at least 1 dose of trial medication in Part B.
Arm/Group | Afatinib Monotherapy (Part A)
Number analyzed (Participants) | 1154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 741
  >=65 years | 413
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 654
  Male | 500
Race/Ethnicity, Customized [Number; unit: Participants]
  Eastern Asian | 491
  Caucasian | 459
  Other | 29
  Unknown | 175
Baseline Eastern Cooperative Oncology Group (ECOG) performance score [Number; unit: Participants] — Subjects were graded based on following ECOG PS grade criteria: Grade 0: Fully active, able to carry on all pre-disease performance without restriction. Grade 1: Restricted in physically strenuous activity but ambulatory & able to carry out work of a light nature. Grade 2: Ambulatory & capable of all selfcare but unable to carry out any work activities. Up & about more than 50% of waking hours. Grade 3: Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours. Grade 4: Completely disabled. Totally confined to bed or chair. Grade 5: Dead.
  Participants
    0 | 341
    1 | 691
    2 | 122
Smoking history [Number; unit: Participants]
  Never smoked | 615
  <15 pack years & stopped >1 year before diagnosis | 132
  Other current or ex-smoker | 407
Histologic classification [Number; unit: Participants]
  Adenocarcinoma | 985
  Squamous | 90
  Other | 78
  Missing | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (Part B)
Description: Progression free survival (PFS) time as determined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 from day of randomization until disease progression or death for patients randomised to combination therapy with afatinib plus paclitaxel or to investigator's choice of chemotherapy.
  Median was calculated from the Kaplan-Meier curve.
Time Frame: From randomization until disease progression or death; Up to 32 months
Population: Randomised Set: This analysis set consist of all randomised patients irrespective of whether treated or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Number analyzed (Participants) | 138 | 68
Months | 5.55 [5.06 to 6.31] | 2.89 [1.87 to 3.94]
Statistical Analysis 1: Comparison: Afatinib Plus Paclitaxel (Part B) vs Investigators Choice of Chemotherapy (Part B); Hazard ratio is calculated from Cox proportional hazard model with treatment as the only factor, stratified by gender and maximum duration of erlotinib or gefitinib (<6 months vs >=6 months); Test type: Superiority or Other; p = 0.0030, stratified log-rank test — P-value is calculated from two-sided stratified log-rank test; Cox Proportional Hazard = 0.61, 95% CI 2-sided [0.44 to 0.85]

2. Secondary Outcome: Progression Free Survival (Part A)
Description: Progression free survival (PFS) as determined by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 for Part A.
  Median was calculated from the Kaplan-Meier curve.
Time Frame: From first dose administration until disease progression or death; Up to 51 months
Population: Treated set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib Monotherapy (Part A)
Number analyzed (Participants) | 1154
Months | 3.15 [2.83 to 3.71]

3. Secondary Outcome: Overall Survival (Part B)
Description: Overall survival (OS) as determined by the time from randomization to death in part B.
  Median was calculated from the Kaplan-Meier curve.
Time Frame: From randomization until death; Up to 32 months
Population: Randomised Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Number analyzed (Participants) | 138 | 68
Months | 12.25 [10.91 to 14.88] | 13.08 [9.86 to 15.64]
Statistical Analysis 1: Comparison: Afatinib Plus Paclitaxel (Part B) vs Investigators Choice of Chemotherapy (Part B); Hazard ratio was calculated from Cox proportional hazard model with treatment as the only factor, stratified by gender and maximum duration of erlotinib or gefitinib (<6 months vs >=6 months); Test type: Superiority or Other; p = 0.7905, Stratified log-rank test; P-value is calculated from two-sided stratified log-rank test; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.76 to 1.44]

4. Secondary Outcome: Objective Response (Part A)
Description: Objective response defined as the best overall response of complete response [CR]: disappearance of all target lesion & partial response [PR]: ≥30% decrease in the sum of the longest diameter of target lesions , taking as reference the baseline sum longest diameter of Afatinib monotherapy according to RECIST 1.1 for Part A.
Time Frame: Post baseline tumour-imaging was performed at every 6 weeks thereafter until disease progression; upto 51 months
Population: Treated set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Monotherapy (Part A)
Number analyzed (Participants) | 1154
Percentage of participants | 8.5 [6.9 to 10.3]

5. Secondary Outcome: Objective Response (Part B)
Description: Objective response (CR, PR) of Afatinib/paclitaxel combination therapy and comparator chemotherapy in Part B after progression in Part A according to RECIST 1.1 .
Time Frame: Post baseline tumour-imaging was performed at every 8 weeks thereafter until disease progression; up to 32 Months
Population: Randomized Set
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Number analyzed (Participants) | 138 | 68
Percentage of participants | 31.2 [23.6 to 39.6] | 13.2 [6.2 to 23.6]
Statistical Analysis 1: Comparison: Afatinib Plus Paclitaxel (Part B) vs Investigators Choice of Chemotherapy (Part B); Odds ratio, 95% Confidence Interval (CI) and p-value (two-sided) from logistic regression stratified for maximum treatment duration of prior erlotinib or gefitinib (>=6 months vs <6 months) and gender; Test type: Superiority or Other; p = 0.0065, Regression, Logistic; Odds Ratio (OR) = 2.980, 95% CI 2-sided [1.357 to 6.543]

6. Secondary Outcome: Intensity and Incidence of Adverse Events (AEs) for Part A & Part B.
Description: Safety of Afatinib as indicated by intensity and incidence of adverse events, graded according to United States National Cancer Institute Common terminology Criteria for Adverse Events (US NCI CTCAE) Version 3.0 both for Part A and Part B. The CTCAE grades are: 1 (mild AE), 2 (moderate AE), 3 (severe AE), 4 (life-threatening or disabling AE), 5 (death related to AE).
Time Frame: From first administration of treatment until 28 days after last drug administration, up to 51 Months (Part A) and from randomization until 28 days after last drug administration of Trial medication, up to 32 Months (Part B)
Population: Treated Set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib Monotherapy (Part A) | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Number analyzed (Participants) | 1154 | 134 | 60
Percentage of participants
  Grade 1 | 8.6 | 4.5 | 8.3
  Grade 2 | 28.0 | 26.1 | 26.7
  Grade 3 | 41.1 | 44.0 | 38.3
  Grade 4 | 4.9 | 9.7 | 6.7
  Grade 5 | 16.6 | 12.7 | 6.7

ADVERSE EVENTS:
Time Frame: From first administration of treatment until 28 days after last drug administration, upto 51 Months (Part A) and from randomization until 28 days after last drug administration of Trial medication, upto 32 Months (Part B).
Description: Part A-events that started within the period defined by the first administration of afatinib until randomization into Part B or 28 days after the last administration of afatinib, whichever occurred first. Part B-events that started within the period from randomization through 28 days after the last administration of trial medication.
Arm/Group | Afatinib Monotherapy (Part A) | Afatinib Plus Paclitaxel (Part B) | Investigators Choice of Chemotherapy (Part B)
Serious Adverse Events (participants affected / at risk) | 471/1154 | 54/134 | 19/60
Other Adverse Events (participants affected / at risk) | 1129/1154 | 128/134 | 50/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Monotherapy (Part A) (N=1154) | Afatinib Plus Paclitaxel (Part B) (N=134) | Investigators Choice of Chemotherapy (Part B) (N=60)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 2 | 1
Ascites (Gastrointestinal disorders) | 4 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 59 | 6 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 18 | 1 | 0
Adverse drug reaction (General disorders) | 0 | 1 | 0
Asthenia (General disorders) | 8 | 1 | 0
Chest pain (General disorders) | 8 | 1 | 1
Extravasation (General disorders) | 0 | 0 | 1
General physical health deterioration (General disorders) | 45 | 7 | 1
Pyrexia (General disorders) | 9 | 1 | 1
Bacterial infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 5 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 42 | 4 | 3
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 5 | 3 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Biopsy lymph gland abnormal (Investigations) | 0 | 1 | 0
Gene mutation identification test (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 0 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 12 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 15 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 46 | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 3 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 19 | 2 | 2
Pericarditis malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 3 | 1 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 1
Seizure (Nervous system disorders) | 6 | 1 | 1
Completed suicide (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 9 | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 67 | 5 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7 | 1 | 0
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 49 | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 17 | 4 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 13 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Shock (Vascular disorders) | 2 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 2 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 3 | 0 | 0
Pericardial effusion (Cardiac disorders) | 5 | 0 | 0
Tachycardia (Cardiac disorders) | 2 | 0 | 0
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal hypomotility (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 2 | 0 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Jejunal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting projectile (Gastrointestinal disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 1 | 0 | 0
Death (General disorders) | 5 | 0 | 0
Fatigue (General disorders) | 4 | 0 | 0
Gravitational oedema (General disorders) | 1 | 0 | 0
Hyperthermia (General disorders) | 1 | 0 | 0
Local swelling (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Mucosal inflammation (General disorders) | 4 | 0 | 0
Multi-organ failure (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0
Pain (General disorders) | 5 | 0 | 0
Performance status decreased (General disorders) | 2 | 0 | 0
Sudden death (General disorders) | 4 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Aspergillus infection (Infections and infestations) | 1 | 0 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 0
Device related infection (Infections and infestations) | 3 | 0 | 0
Endocarditis (Infections and infestations) | 1 | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 0
Escherichia sepsis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 2 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0
Lung abscess (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 11 | 0 | 0
Lymphangitis (Infections and infestations) | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0
Peritonitis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 5 | 0 | 0
Septic shock (Infections and infestations) | 5 | 0 | 0
Skin bacterial infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 1 | 0 | 0
Staphylococcus test positive (Investigations) | 1 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant neoplasm of pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Brain oedema (Nervous system disorders) | 3 | 0 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 4 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 5 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 2 | 0 | 0
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Reversible ischaemic neurological deficit (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 2 | 0 | 0
Spinal cord compression (Nervous system disorders) | 4 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Anuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Pleural fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thoracic haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Lung transplant (Surgical and medical procedures) | 1 | 0 | 0
Partial lung resection (Surgical and medical procedures) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 6 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0
Neurogenic shock (Vascular disorders) | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib Monotherapy (Part A) (N=1154) | Afatinib Plus Paclitaxel (Part B) (N=134) | Investigators Choice of Chemotherapy (Part B) (N=60)
Anaemia (Blood and lymphatic system disorders) | 80 | 33 | 6
Leukopenia (Blood and lymphatic system disorders) | 5 | 20 | 7
Neutropenia (Blood and lymphatic system disorders) | 7 | 26 | 8
Abdominal pain (Gastrointestinal disorders) | 90 | 11 | 4
Abdominal pain upper (Gastrointestinal disorders) | 65 | 19 | 4
Constipation (Gastrointestinal disorders) | 85 | 22 | 10
Diarrhoea (Gastrointestinal disorders) | 964 | 72 | 4
Nausea (Gastrointestinal disorders) | 252 | 28 | 14
Stomatitis (Gastrointestinal disorders) | 303 | 14 | 2
Vomiting (Gastrointestinal disorders) | 211 | 31 | 4
Asthenia (General disorders) | 200 | 47 | 18
Chest pain (General disorders) | 82 | 9 | 2
Fatigue (General disorders) | 136 | 32 | 10
Mucosal inflammation (General disorders) | 200 | 13 | 0
Oedema peripheral (General disorders) | 57 | 12 | 2
Pyrexia (General disorders) | 82 | 18 | 7
Bronchitis (Infections and infestations) | 21 | 7 | 2
Conjunctivitis (Infections and infestations) | 79 | 12 | 0
Nasopharyngitis (Infections and infestations) | 35 | 10 | 2
Paronychia (Infections and infestations) | 342 | 23 | 0
Pneumonia (Infections and infestations) | 68 | 8 | 1
Rhinitis (Infections and infestations) | 54 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 32 | 7 | 1
Urinary tract infection (Infections and infestations) | 62 | 14 | 1
Alanine aminotransferase increased (Investigations) | 28 | 8 | 2
Haemoglobin decreased (Investigations) | 11 | 7 | 0
Weight decreased (Investigations) | 132 | 16 | 3
Decreased appetite (Metabolism and nutrition disorders) | 304 | 37 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 51 | 12 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 46 | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 94 | 8 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 48 | 8 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 17 | 10 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 | 8 | 5
Dizziness (Nervous system disorders) | 60 | 13 | 4
Dysgeusia (Nervous system disorders) | 25 | 7 | 4
Headache (Nervous system disorders) | 56 | 16 | 6
Hypoaesthesia (Nervous system disorders) | 6 | 9 | 5
Neuropathy peripheral (Nervous system disorders) | 8 | 16 | 7
Paraesthesia (Nervous system disorders) | 25 | 13 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 8 | 2
Insomnia (Psychiatric disorders) | 39 | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 194 | 32 | 13
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 36 | 7 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 194 | 34 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 151 | 19 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 10 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 47 | 6 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 39 | 47 | 10
Nail disorder (Skin and subcutaneous tissue disorders) | 41 | 9 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 179 | 13 | 3
Rash (Skin and subcutaneous tissue disorders) | 629 | 30 | 7
Skin fissures (Skin and subcutaneous tissue disorders) | 101 | 10 | 1
Mouth ulceration (Gastrointestinal disorders) | 91 | 2 | 0
Folliculitis (Infections and infestations) | 86 | 5 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 61 | 6 | 4
Acne (Skin and subcutaneous tissue disorders) | 87 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 164 | 6 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 71 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.